CLINICAL TRIAL: NCT04476069
Title: Effect of Preoperative Administration of Ibuprofen in Children Undergoing Extraction for Reducing Postoperative Pain: A Double-blind Randomized Controlled Clinical Trial
Brief Title: Ibuprofen as a Pain Management in Pediatric Dentistry
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Princess Nourah Bint Abdulrahman University (Other)
Responsible Party: Principal Investigator, Abeer ali alshami, Assistant professor / Consultant in Pediatric dentistry, Princess Nourah Bint Abdulrahman University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: H-01-R059
Record Dates: First submitted 2020-07-09; First posted 2020-07-17 (Actual); Last update posted 2020-07-17 (Actual); Status verified 2020-07

CONDITIONS: Pain Management
MeSH Terms: conditions — Agnosia | interventions — Ibuprofen

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind, placebo-controlled clinical trial
Who Masked: Participant, Care Provider, Investigator
Masking Description: a professional research coordinator is hired to develop blinded materials. A list of identification numbers will be created, and each number will randomly be assigned to either Group A (receive ibuprofen prior to extraction) or Group B (receive placebo prior to extraction, as a control). Only the RC will know the assignment of the numbers to groups. Blinded medications will be developed and labelled according to the identification (ID) numbers.
  Once participants undergo consent, they will be assigned an ID number which placed them in a randomized group. The clinician will the medication associated with the participant's ID number prior to extraction.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ibuprofen (Experimental): 30 minutes before extraction, once/day orally
  Interventions: Drug: IBUPROFEN
- Placebo (Placebo Comparator): 30 minutes before extraction, once/day orally
  Interventions: Drug: IBUPROFEN

INTERVENTIONS:
Drug: IBUPROFEN — given to children 30 minutes before extraction / orally for one time only

SUMMARY:
Abstract Introduction: Administration of non-steroidal anti-inflammatory drugs (NSAIDs) before tooth extraction may reduce post-surgical pain, but there is a lack of research.

Aims: To compare pain and anxiety in pediatric tooth extraction patients receiving a preoperative NSAID vs. placebo.

Design: Randomized, double-blind, placebo-controlled clinical trial. Setting: Princess Nourah Bint Abdulrahman University's (PNU's) dental clinic in Riyadh, Saudi Arabia.

Materials and Methods: Eligible pediatric tooth extraction patients were randomized to Group A, which received NSAID preoperatively, or Group B, which received placebo.

Interventions: A research coordinator (RC) measured participants prior to extraction, and 3- and 24-hours post-extraction.

Main Outcome Methods: The Wong-Baker FACES scale (WBFS) and the Modified Child Dental Anxiety Scale - Faces (MCDASf).

DETAILED DESCRIPTION:
Aims The aim of this study was to compare the post-operative pain and anxiety experience of pediatric tooth extraction patients who receive a preoperative NSAID with those who receive a placebo in order to evaluate the impact of preoperative NSAID administration on post-surgical pain and anxiety.

Design This was a randomized, double-blind, placebo-controlled clinical trial. Setting This study was conducted at Princess Nourah Bint Abdulrahman University's (PNU's) dental clinic in Riyadh, Saudi Arabia.

Materials and Methods Participants Pediatric patients were referred to the study by clinicians at the PNU clinic. Inclusion criteria included: child must have been age five through 13; child must be undergoing a simple extraction under local anesthesia of one or more symptomatic primary molars including teeth with pathology such as abscess, cyst, and internal resorption; parent must provide consent and the child provide assent; child must not have any systematic disease, child must not be taking any medication that interacts with ibuprofen (the NSAID used in this study), and child must be cooperative. Children were excluded for known allergy or having ever had an allergic reaction to ibuprofen; taking antibiotics or other medications; having special needs due to a physical or mental disability; having been given an analgesic prior to appointment by guardian; or being treated for an emergency medical condition (e.g., cellulitis). This study was reviewed and approved by the PNU Research Ethics Board (REB).

Records of potential participants were reviewed prior to inviting them into study participation so that they were already screened for inclusion and exclusion criteria and they were known to qualify. This was a clinical study, and recruitment was limited to participants who qualified, although a total sample size of 60 was thought to be possible and so was targeted.

Randomization, Blinding, and Baseline Data Collection To facilitate double-blinding, a professional research coordinator (RC) was hired to develop blinded materials. A list of identification numbers was created and each number was randomly assigned to either Group A (receive ibuprofen prior to extraction) or Group B (receive placebo prior to extraction, as a control). Only the RC knew the assignment of the numbers to groups. Blinded medications were developed and labeled according to the identification (ID) numbers.

Once participants underwent consent, they were assigned an ID number which placed them in a randomized group. The clinician used the medication associated with the participant's ID number prior to extraction. At this point, baseline data was gathered, which included the following variables: patient gender, patient age, anesthesia technique used (infiltration for upper mouth extractions, and nerve block for lower mouth extractions), number of teeth being extracted, baseline self-reported pain measurement, and baseline self-reported anxiety measurement.

Interventions Administration of Study Drug Once placed in a randomization group, the study drug was administered. Those randomized to Group A (active) received the NSAID in the study, which was oral commercially-available Nurfen® syrup containing the NSAID ibuprofen. Between 7.5 to 15 ml/kg was administered, depending on the child's age. Those randomized to Group B (control) were given a colored, flavored solution as a placebo.

Tooth Extraction After administration of the study drug and baseline data collection, the treating clinicians (n=6) followed a standard protocol for the study. Clinicians had 1 to 5 years of experience. No formal calibration was done, and behavioral management techniques were included in the standard protocol. They reviewed the participant's medical and dental histories and noted any allergies. After a thorough clinical and radiographic examination, they applied topical anesthesia, then administered local anesthesia with dosage appropriate to the patient's age and weight (Lidocaine 2% with epinephrine 1:100,000). After local anesthesia, the efficacy of the anesthesia was tested subjectively and objectively, then pediatric forceps were used for the extraction(s). This was followed by the application of a gauze pressure pack, and verbal and written post-extraction instructions were provided to the child and parent.

Main Outcome Methods Data Collection Two instruments were used for outcome measurement: the Wong-Baker FACES scale (WBFS) for pain perception, and the Modified Child Dental Anxiety Scale - Faces (MCDASf) for anxiety. Both the WBFS and MCDASf were administered at baseline (immediately after consent), and at 3- and 24-hours post-extraction. It was estimated that 3-hours post-extraction, local analgesic would have worn off and pain would typically be at its peak.

The baseline measurements were done in person by the RC, and both the 3- and 24-hour follow-up measurements were conducted by the RC by phone. As both WBFS and MCDASf are visual scales, forms were provided to the parent at the appointment which were then completed with the child during the follow-up calls and sent to the RC in the mail. During the follow-up phone calls, the researcher would talk on the phone to the parent, and coach them to ask the child the questions and have the child answer them by pointing to the visual scale. The parent would the relay the child's answer to the researcher for the record.

Measurements Intended for pediatrics patients, the WBFS has patients assign a score of 0, 2, 4, 6, 8, and 10 to indicate their level of perceived pain.

The MCDASf scale was developed and validated to measure dental-related anxiety in children about eight different topics; only "How do you feel about having a tooth taken out?" was asked in this study. Respondents assign a score between 1 and 5 corresponding to their level of anxiety about the topic .

ELIGIBILITY:
Inclusion Criteria:

1. child must be undergoing a simple extraction under local anesthesia of one or more symptomatic primary molars including teeth with pathology such as abscess, cyst, and internal resorption
2. parent must provide consent and the child provide assent
3. must not have any systematic disease
4. must not be taking any medication that interacts with ibuprofen (the NSAID used in this study)
5. must be cooperative

   * Excluded Criteria Children were excluded for

1-known allergy 2-having ever had an allergic reaction to ibuprofen 3- taking antibiotics or other medications 4-special needs due to a physical or mental disability 5-been given an analgesic prior to appointment by the guardian; 6-being treated for an emergency medical condition (e.g., cellulitis).

Ages: 5 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 56 (Actual)
Dates: Start 2019-01-10 (Actual); Primary Completion 2019-03-28 (Actual); Study Completion 2019-05-30 (Actual)

PRIMARY OUTCOMES:
To compare pain and anxiety in pediatric tooth extraction patients receiving a preoperative NSAID vs. placebo | First 24 hours after drug administration
  Main Outcome Methods: measurement of the Wong Baker Faces (WBFS) scale has been used and patients assign a score of 0, 2, 4, 6, 8, and 10 to indicate their level of perceived pain.
  Score 10 is the highest level of pain

CONTACTS AND LOCATIONS:
Overall Officials: Abeer A Alshami, PhD, Principal Investigator — Princess Noura Bint Abdulrhman University
Locations (1):
- College of Dentistry /Princess Nourah Bint Abdulrhman University, Riyadh, Saudi Arabia

IPD SHARING:
Plan to Share IPD: Yes
All of the individual participant data collected during the trial, after deidentification.
Supporting Information: Study Protocol
Time Frame: Immediately following publication. No end date.
Access Criteria: Anyone who wishes to access the data.

REFERENCES:
- [Result] Ashley PF, Parekh S, Moles DR, Anand P, MacDonald LC. Preoperative analgesics for additional pain relief in children and adolescents having dental treatment. Cochrane Database Syst Rev. 2016 Aug 8;2016(8):CD008392. doi: 10.1002/14651858.CD008392.pub3. PMID 27501304
- [Result] Al-Namankany A, de Souza M, Ashley P. Evidence-based dentistry: analysis of dental anxiety scales for children. Br Dent J. 2012 Mar 9;212(5):219-22. doi: 10.1038/sj.bdj.2012.174. PMID 22402535